CLINICAL TRIAL: NCT01748591
Title: A Study of PICOPREP in Patients Needing to Clean the Bowel Prior to X-ray Examination, Endoscopy or Surgery
Brief Title: Monitoring of Safety and Tolerance of PICOPREP in Clinical Practice
Status: Terminated | Type: Observational
Why Stopped: Terminated due to problems enrolling adequate number of patients.
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: 000062
Record Dates: First submitted 2012-11-09; First posted 2012-12-12 (Estimated); Last update posted 2015-12-22 (Estimated); Status verified 2015-12

CONDITIONS: Bowel Cleanliness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- PICOPREP treatment: PICOPREP powder for oral solution according to standard clinical practice

SUMMARY:
A Confirmation of Safety, Tolerance and Efficacy of PICOPREP in Clinical Practice.

ELIGIBILITY:
Inclusion Criteria:

* Patients eligible for treatment with PICOPREP® for bowel cleansing prior to endoscopic examination or surgery

Exclusion Criteria:

* Patients in which prescription of PICOPREP® is contraindicated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients eligible for endoscopic examination or surgery
Sampling Method: Non-Probability Sample
Enrollment: 3324 (Actual)
Dates: Start 2012-05; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
The Frequency of Adverse Events | 2 days
The Severity of Adverse Events | 2 days

SECONDARY OUTCOMES:
Treatment efficacy measured by assessment of the quality of colon cleaning | 2 days

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals
Locations (22):
- Czechia (22):
  - Nemocnice Rudolfa a Stefanie, Benešov
  - Nemocnice Blansko, Blansko
  - Nemocnice Břeclav, Břeclav
  - Soukrmá ambulance, Česká Lípa
  - Děčínská nemocnice, Děčín
  - Nemocnice Havlíčkův Brod, Havlíčkův Brod
  - Fakultní nemocnice Hradec Králové, Hradec Králové
  - Nemocnice Jablonec, Jablonec nad Nisou
  - Nemocnice Jihlava, Jihlava
  - Privátní GE, Jihlava
  - FN Olomouc, Olomouc
  - FN Bulovka, Prague
  - Privátní GE Praha 4, Prague
  - Sanatorium Sv.Anny, Prague
  - Thomayerova nemocnice, Prague
  - Všeobecná fakutlní nemocnice, Prague
  - Nemocnice Příbram, Příbram
  - Lužická nemocnice, Rumburk
  - Nemocnice Tábor, Tábor
  - Nemocnice Teplice, Teplice
  - Ústecká poliklinika, Ústí nad Labem
  - Nemocnice Znojmo, Znojmo